CLINICAL TRIAL: NCT06963424
Title: Pain Relief and Peripheral Perfusion Index When Local Anesthetics Injected in Different Final Target Area During Lumbar Erector Spinae Block
Brief Title: Pain Relief and and Peripheral Perfusion Index During Erector Spinae Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-02-028
Record Dates: First submitted 2025-04-29; First posted 2025-05-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Block; Block, Fascicular; Spinae
MeSH Terms: conditions — Bites and Stings; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intertransverse ligagment group (Experimental): lumbar ESPB was performed with final target at intertransverse ligament
  Interventions: Procedure: Erector Spinae Plane Block
- transverse process group (Placebo Comparator): lumbar ESPB was performed with final target at transverse process
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — lumbar erectro spinae block

SUMMARY:
The primary endpoint of this study is to compare the pain relief and peripheral perfusion index when local anesthetics injected in different final target area during lumbar erector spinae block The secondary endpoint of this study is to compare the procedure related pain

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. The final target area of ESPB of cervical, thoarcic, and lumbar regiona is transverse process. Once the needle contact the tip of the transverse process, local anesthetics is injected subsequentely. However, contacting the bony structure with the needle can generage procedure related pain. If ESPB can be performed without touching the transverse process, the satisfaction of patient would be increased. Actually, intertransverse ligament, which is visibe by ultrasound, is present between transverse process. Therefore, if local anesthetics is injected after targeting intertransverse ligament, same effect of pain relief with tarting of transverse process of ESPB is uncertain

ELIGIBILITY:
Inclusion Criteria:

* lumbar disc herniation
* lumbar foraminal stenosis
* lumbar central stenosis
* lumbar spondylolisthesis
* numerical rating scale > 4
* back pain functional scale < 45
* duration of pain > 1 mon
* patients who can fully understand all items described in back pain functional scale

Exclusion Criteria:

* Allergy to local anesthetics or contrast medium
* Pregnancy
* Spine deformity
* Prior history of lumbar spine surgery
* No previous lumbar MRI or CT
* Patients with coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale changes among 5 times period | Baseline, 2 weeks, 4 weeks, 8 weeks after the completion of erector spine plane block
  minimum (1) and maximum value (10), lower score means better treatment outcome

SECONDARY OUTCOMES:
back pain functional scale among 3 times period | Baseline, 4 weeks, 8 weeks after the completion of erector spine plane block
  minimum (0) and maximum value (60), higher score means better treatment outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Ji Hee, Daegu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No